CLINICAL TRIAL: NCT01082172
Title: A Pilot Trial to Evaluate the Performance of the TriVascular Thoracic Stent Graft System
Brief Title: South American Thoracic Stent-Graft Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriVascular, Inc. (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 771-0001 TAA Trial
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: thoracic; aortic; aneurysm; TAA
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic Stent Graft (Experimental): Thoracic Stent Graft implanted device
  Interventions: Device: Implant Thoracic Stent Graft

INTERVENTIONS:
Device: Implant Thoracic Stent Graft — Endovascular implant of Thoracic Aortic Aneurysm Stent Graft

SUMMARY:
A prospective, non-randomized multi-center clinical evaluation of the performance of the TriVascular Thoracic Stent Graft System when used in the treatment of subjects with thoracic aortic aneurysms (TAA).

ELIGIBILITY:
Inclusion Criteria:

* The TriVascular Thoracic Stent Graft System is indicated in subjects diagnosed with an aneurysm in the descending thoracic aorta having vascular morphology suitable for endovascular repair, including:

  * Adequate iliac/femoral access compatible with the required delivery systems,
  * Non-aneurysmal aortic segments proximal and distal to the aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Absence of device-related serious adverse events within 30-days of endovascular procedure | 30-Days

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Caolica de Chile, Santiago, Chile